CLINICAL TRIAL: NCT03037905
Title: Effect of the Built Operating Room Environment on Patient Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: STERIS Corporation (Unknown)
Responsible Party: Principal Investigator, Christian Burchill, Nurse Scientist II, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCF15-009
Record Dates: First submitted 2016-09-11; First posted 2017-01-31 (Estimated); Results first posted 2017-11-22 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SignatureSuite OR (Experimental): The intervention is exposure to the operating room environment created by the device SignatureSuite OR Integration System by STERIS Corporation.
  Interventions: Device: SignatureSuite OR Integration System by STERIS Corporation
- Standard OR (No Intervention): Standard operating room without SignatureSuite OR Integration System by STERIS Corporation.

INTERVENTIONS:
Device: SignatureSuite OR Integration System by STERIS Corporation — SignatureSuite OR Integration System by STERIS Corporation is a device that controls audio and visual components of the operating room environment in order to provide a more relaxing and calming operating room environment for patients prior to surgery and on emergence from anesthesia after surgery.
  Other Names: SignatureSuite
  Arms: SignatureSuite OR

SUMMARY:
Anxiety prior to surgery is an expected emotion. Research has not been conducted on methods to reduce anxiety in the operating room itself. STERIS Corporation has developed an automated surgical suite environmental system, called SignatureSuite™, that controls the level of lighting, images on OR monitors, and ambient background audio via preset, computerized automation for use before and after anesthesia. This study aims to determine if this new type of operating room environment decreases anxiety, as measured by patient responses on anxiety visual analog scales, heart rate, systolic blood pressure, and postoperative analgesic use. The proposed study will be a two-arm, randomized controlled trial comparing anxiety levels for patients that have thyroid or parathyroid surgery in the SignatureSuite room at Cleveland Clinic Marymount Hospital versus the standard operating room environment. Randomization will occur at the surgeon level. There will be a maximum 100 patients divided equally between the experimental and control arms of the study.

DETAILED DESCRIPTION:
Problem: Anxiety prior to surgery is an expected emotion. Research has been conducted on methods to reduce anxiety prior to entering the operating room (OR). These studies have involved some form of distraction, almost all finding that some form of distraction prior to entering the OR decreases both physiologic signs and patient reports of anxiety. Very few of these studies have carried the intervention into the OR itself. Steris Corporation has developed an automated surgical suite environmental system, called SignatureSuite™, that controls the level of lighting, images on OR monitors, and ambient background audio via preset, computerized automation for use before and after anesthesia. The research question is: What is the effect of the SignatureSuite OR environment on patient anxiety and analgesic use? Study methods: The proposed study will be a two arm randomized controlled trial. Randomization will occur at the surgeon level, based on SignatureSuite operating room environment (experimental group) versus a standard Marymount Hospital operating room environment (control group).

Data collection: The study will take place in the perioperative department of Cleveland Clinic's Marymount Hospital. Patient anxiety will be measured before and after surgery using an anxiety visual analog scale (VAS). Data about patient characteristics will be retrieved retrospectively by chart review. The effect of SignatureSuite on OR time will also be determined.

Sample characteristics: The patient sample will comprise patients undergoing thyroid and/or parathyroid surgery at Cleveland Clinic Marymount Hospital.

Sample size: 40 subjects per group will provide adequate power to detect large effect sizes (0.80) and is feasible in a reasonable period of time.

ELIGIBILITY:
Inclusion Criteria:

* able to read and understand English;
* presentation for thyroid and/or parathyroid surgery at Marymount Hospital;
* visual capacity to complete the VAS

Exclusion Criteria:

* history of documented anxiety/depression disorder
* currently taking medications for depression/anxiety
* currently taking anticonvulsant medication and/or gamma-Aminobutyric acid analogs
* unable to read and understand English
* dementia
* vision loss making it impossible to complete the anxiety visual analog scale
* currently taking beta-blockers
* surgeon refusal for patient participation
* intra-operative emergency, such as cardiac incident requiring resuscitation or stabilizing medications, unplanned extubation, or early emergence from anesthesia
* other patient-related reasons that would affect eligibility to participate.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian N Burchill, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Marymount Hospital, Garfield Heights, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No data to be shared

RESULTS

PARTICIPANT FLOW:
Groups:
- SignatureSuite OR: Patients who's surgeon has been randomized into the SignatureSuite operating room. The intervention is the unique operating room environment created by the product.
  SignatureSuite™ OR Integration System by STERIS Corporation: SignatureSuite™ OR Integration System by STERIS Corporation is a product that includes software to control the audio and visual components of the operating room in order to provide a more relaxed and calming environment for patients prior to their surgery. It automatically dims lights, plays pleasant music or sounds of nature over the in-room speakers, and provides scenes of nature on video screens stationed in viewing range of the patient. As anesthesia is administered to the patient, the system automatically adjusts the light and sound systems to come up to surgeon-preferred preset stations. The process happens in reverse as the patient emerges from general anesthesia so that they awaken in the same environment as when they arrived in the OR.
- Standard OR: Patients who's surgeon has been randomized into the standard operating room.
Period: Overall Study
Arm/Group | SignatureSuite OR | Standard OR
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Thyroid surgery cases
Groups:
- Total: Total of all reporting groups
Arm/Group | SignatureSuite OR | Standard OR | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (14.3) | 53.3 (14.3) | 52.5 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 43 | 84
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 49 | 48 | 97
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 12 | 15
  White | 41 | 36 | 77
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 3 | 0 | 3
Surgical site [Count of Participants; unit: Participants]
  Parathyroid | 16 | 22 | 38
  Thyroid | 34 | 28 | 62
Kindler Preoperative Anxiety Scale Total Score [Median (Inter-Quartile Range); unit: units on a scale] — The Kindler preoperative anxiety scale quantifies 10 factors that cause preoperative anxiety. Each factor is measured on a 100 millimeter line with anchors "No anxiety" to "The most anxiety I can imagine." Participants make a mark across the line to represent their current state on each factor. A millimeter ruler is used to measure from left to right with the number of millimeters recorded where the mark crosses the line, minimum score is 0 and maximum score is 100. Higher number means more anxiety. The average of the scores represents the total preoperative anxiety score.
  units on a scale | 29.8 [15.8 to 55.2] | 26.6 [8.6 to 44.1] | 28.9 [10.3 to 47.9]
Past medical history diagnosis groups [Number; unit: participants]
  cardiovascular/respiratory | 13 | 19 | 32
  Other | 15 | 19 | 34
  endocrine | 49 | 48 | 97
  gastrointestinal/genitourinary | 20 | 18 | 38
  neuromuscular | 16 | 25 | 41
Preoperative anxiety visual analog scale [Mean (Standard Deviation); unit: units on a scale] — The preoperative anxiety scale quantifies preoperative anxiety. It is measured on a 100 millimeter line with anchors "No anxiety" to "The most anxiety I can imagine." Participants make a mark across the line to represent their current state of preoperative anxiety. A millimeter ruler is used to measure from left to right with the number of millimeters recorded where the mark crosses the line, minimum score is 0 and maximum score is 100. Higher number means more anxiety.
  units on a scale | 36.3 (27.9) | 32.0 (28.9) | 34.13 (28.4)
Preoperative systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 137.50 (17.4) | 142.6 (19.8) | 140.0 (18.7)
Preoperative heart rate [Mean (Standard Deviation); unit: beats per minute] | 77.9 (12.7) | 78.8 (15.3) | 78.4 (14.0)

OUTCOME MEASURES:

1. Primary Outcome: Change (Difference) in Anxiety
Description: Change (difference) in anxiety level as measured by a 100 millimeter line visual analog scale from baseline (pre-operative) to arrival in post anesthesia care unit (post-operative).The anxiety visual analog scale quantifies current state of anxiety. It is measured on a 100 millimeter line with anchors "No anxiety" to "The most anxiety I can imagine." Participants make a mark across the line to represent their current state of anxiety. A millimeter ruler is used to measure from left to right with the number of millimeters recorded where the mark crosses the line, minimum score is 0 and maximum score is 100. Higher number means more anxiety.
Time Frame: Pre-operatively to post-operatively
Population: thyroid and/or parathyroid surgery patients
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SignatureSuite OR | Standard OR
Number analyzed (Participants) | 50 | 50
units on a scale | -24.4 [-31.7 to -17.0] | -17.6 [-25.1 to -10.2]
Statistical Analysis 1: Comparison: SignatureSuite OR vs Standard OR; Test type: Superiority; p = 0.20, Mixed Models Analysis; Mean Difference (Final Values) = -6.7, 95% CI 2-sided [-17.1 to 3.7]

2. Secondary Outcome: Difference Between Pre-operative Systolic Blood Pressure and a Mean of 3 Post-operative Systolic Blood Pressures
Description: Difference between pre-operative systolic blood pressure and a mean of 3 post-operative systolic blood pressures assessed at 15, 30 and 45 minutes after placement in post-anesthesia care unit
Time Frame: Pre-operative to post-operative
Population: Patients undergoing thyroid and/or parathyroid surgery
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | SignatureSuite OR | Standard OR
Number analyzed (Participants) | 50 | 50
mm Hg | -4.2 [-9.8 to 1.4] | -6.4 [-12.3 to -0.5]
Statistical Analysis 1: Comparison: SignatureSuite OR vs Standard OR; Test type: Superiority; p = 0.60, Mixed Models Analysis; Mean Difference (Final Values) = 2.2, 95% CI 2-sided [-5.9 to 10.3]

3. Secondary Outcome: Difference Between Pre-operative Heart Rate and a Mean of 3 Post-operative Heart Rates
Description: Difference between pre-operative heart rate and a mean of 3 post-operative heart rates assessed at 15, 30 and 45 minutes after placement in post-anesthesia care unit
Time Frame: Pre-operative to post-operative
Population: Patients undergoing thyroid and/or parathyroid surgery
Measure: Mean (95% Confidence Interval); unit: beats per minute
Arm/Group | SignatureSuite OR | Standard OR
Number analyzed (Participants) | 50 | 50
beats per minute | 3.1 [-1.3 to 7.5] | 4.1 [-0.2 to 8.3]
Statistical Analysis 1: Comparison: SignatureSuite OR vs Standard OR; Test type: Superiority; p = .76, Mixed Models Analysis; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-7.0 to 5.1]

4. Other Pre Specified Outcome: Analgesic Use
Description: Number of people requiring analgesia in the post-anesthesia care unit
Time Frame: Postoperatively
Population: Patients that have undergone thyroid and/or parathyroid surgery
Measure: Count of Participants; unit: Participants
Arm/Group | SignatureSuite OR | Standard OR
Number analyzed (Participants) | 50 | 50
Participants | 9 | 10
Statistical Analysis 1: Comparison: SignatureSuite OR vs Standard OR; Test type: Superiority; p = .83, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Postoperatively until discharged from the post-anesthesia care unit.
Arm/Group | SignatureSuite OR | Standard OR
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
Study was conducted at one community hospital in Northeast Ohio. Study population limited to patients having thyroid or parathyroid surgery. Low dose anxiolytic given intravenously in the preoperative holding area prior to being moved to the OR.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No